CLINICAL TRIAL: NCT02819466
Title: Visualization of the Stomach During Fasting and Measurement of Intragastric Volume After Ingestion of Fluid: Feasibility and Application of Three Dimensional Ultrasound in Healthy Subjects. ECHO3DGASTRIQUE Study
Brief Title: Visualization of the Stomach During Fasting and Measurement of Intragastric Volume After Ingestion of Fluid: Feasibility and Application of Three Dimensional Ultrasound in Healthy Subjects
Acronym: ECHO3DGASTRIQ
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2012_843_0027
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Echocardiography, Three-Dimensional
Keywords: intragastric volume; stomach; fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- volunteers: Healthy volunteers over the age of 18 years employed by Amiens University Hospital 3D echography
  Interventions: Device: 3D echography

INTERVENTIONS:
Device: 3D echography — ultrasound visualization of the stomach in fasting patients.

SUMMARY:
Aspiration pneumonia is a dreaded complication of anaesthesia because of its prevalence (1/3,886 cases in elective anaesthesia and 1/895 cases in emergency settings) and its high morbidity and mortality (3 to 9%). This chemical and/or infectious pneumonia is secondary to passage of the gastric contents into the unprotected upper airways during general anaesthesia. The prognosis depends on three factors: the presence of food debris, and the acidity and volume of the gastric contents. To prevent this complication, the French society of anaesthesia and intensive care recommends preoperative fasting rules and, in patients presenting risk factors for aspiration, the use of antacids and rapid sequence intubation. This preventive strategy is associated with certain adverse events: deferred operative procedures, discomfort and hypoglycaemia secondary to fasting, more frequent anaphylactic complications, and memory of anaesthetic induction.

Over recent years, ultrasound has become more widely used by anaesthetists for local anaesthesia, vascular catheterization, haemodynamic monitoring and, more recently, 2D ultrasound estimation of intragastric volume. However, 2D ultrasound estimation of intragastric volume presents several limitations: because of the complex shape of the stomach, this technique requires a long learning curve and the measured volume is poorly correlated with reference techniques (MRI and 99Tc scintigraphy). Two studies have recently measured intragastric volume by three dimensional ultrasound with promising results.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers over the age of 18 years employed by Amiens University Hospital and covered by French national health insurance.
* Fasting (last meal > 6 hours and last drink of water, tea or coffee > 2 hours)
* Signature of the free and informed written consent form.

Exclusion Criteria:

* Pregnant woman.
* Presence of diseases or treatments that alter (slow or accelerate) gastric emptying.
* Presence of swallowing disorders.
* History of gastric or supramesocolic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers fasting
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
success rate of ultrasound visualization of the stomach while fasting | Day 0
  success rate of ultrasound visualization of the stomach while fasting

SECONDARY OUTCOMES:
ultrasound visualization of the fasting stomach learning curve | Day 0
  ultrasound visualization of the fasting stomach learning curve for each investigator
measured difference of antral surface area | Day 0
  antral surface area after ingestion of fluid - fasting antral surface area
absolute error of the volume measured | Day 0
  ingested volume - intragastric volume variation
relative error of the volume measured | Day 0
  (absolute error / ingested volume) * 100

CONTACTS AND LOCATIONS:
Overall Officials: Edouard SECQ, PhD, Principal Investigator — CHU Amiens; Emmanuel LORNE, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France